CLINICAL TRIAL: NCT07022106
Title: Comparison of Myofascial Release and Kinesiotaping Techniques in the Management of Primary Dysmenorrhea
Brief Title: Comparison of Different Physiotherapy Techniques in Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Salma Abdelzaher, Physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: E-10840098-202.3.02-582
Record Dates: First submitted 2025-05-30; First posted 2025-06-15 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Dysmenorrhea Primary
Keywords: primary dysmenorrhea; kinesiotape; myofascial release; pain
MeSH Terms: conditions — Pain | interventions — Myofascial Release Therapy; Population Groups; Athletic Tape

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesiotape (KT) Group (Experimental): Participants in this arm will receive Kinesio Taping applied to the lower abdomen and lumbar region using a 3-Tape Sensory Modulation Technique to modulate pain and fascial tension.
  Interventions: Other: Kinesiotape (KT) Group
- Myofascial Release Therapy (MRT) Group (Experimental): Participants in this arm will receive a single session of myofascial release technique (MRT) which is a type of massage that will target anterolateral abdominal wall, including Camper and Scarpa fascia, as well as the deeper layers, including transversals fascia and the thoracolumbar fascia to release the fascial restrictions.
  Interventions: Other: Myofascial Release Therapy (MRT) Group

INTERVENTIONS:
Other: Myofascial Release Therapy (MRT) Group — Myofascial Release Therapy (MRT) involves hands-on palpation to detect fascial restrictions, followed by 60-90 seconds of sustained pressure to release tension. In the supine position, the target areas include the superficial fascia, transversalis fascia, and extraperitoneal fascia, while in the prone position, the focus shifts to the thoracolumbar fascia and the erector spinae complex. This technique aims to restore mobility and reduce restrictions within the fascial system.
  Frequency: Each patient will recieve a single session at their most painful day from this intervention.
  Arms: Myofascial Release Therapy (MRT) Group
Other: Kinesiotape (KT) Group — Kinesio Taping (KT) Intervention
  Description:
  Participants will receive a standardized 3-tape sensory modulation technique using Kinesiotape, applied to the abdomen and sacrum to target fascial tension and visceral pain in primary dysmenorrhea.
  Procedure:
  Abdominal Application (Two Tapes, 0% Stretch):
  Horizontal Tape: Placed between the iliac crests (lower abdomen) to reduce fascial tension.
  Vertical Tape: Applied from the navel to the pubic symphysis to modulate visceral pain signaling.
  Sacral Application (One Tape, 15-25% Stretch):
  Horizontal Tape: Anchored across the S2-S4 vertebrae (at PSIS level) to activate the pain-gating mechanism via cutaneous-visceral reflexes.
  Frequency/Duration:
  Each participant will receive a single session at their most painful day from this intervention
  Arms: Kinesiotape (KT) Group

SUMMARY:
This study is investigating the effects of myofascial release technique & kinesiotape in managing dysmenorrhea

DETAILED DESCRIPTION:
Dysmenorrhea is a common gynecological disorder characterized by painful menstruation manifested by severe cramps in the lower abdomen. Recent epidemiological studies indicate a global prevalence of 50-90% among women (10-20% with severe symptoms); in Türkiye, studies show a prevalence of 75-85%.Dysmenorrhea is divided into two types: primary dysmenorrhea (PD) and secondary dysmenorrhea. PD is painful menstruation without any underlying pathological condition. The main goal of dysmenorrhea treatment is to significantly improve the patient's well-being and quality of life (QoL) by effectively relieving pain and relieving symptoms by targeting physiological mechanisms. There are various physiotherapy methods that can be used to reduce this pain, such as transcutaneous electrical nerve stimulation (TENS), cryotherapy, myofascial release therapy (MRT), and kinesiology taping (KT).

This single-blind randomized controlled trial will investigate the acute therapeutic effects of Myofascial Release Technique (MRT) versus Kinesio Taping (KT) in 46 females aged 18-30 years with PD. Participants will be randomised into Group 1 (MRT; n = 23) or Group 2 (KT; n = 23), receiving a single intervention session during their most painful menstrual day

All participants will be asked to fill out 3 forms, namely a sociodemographic questionnaire covering age, height, BMI, age at menarche and duration of menstruation, a Visual Analog Scale (VAS) to assess pain level and a Patient Reported Outcomes Measurement System (PROMIS-29 Profile v2.0) to measure quality of life (QoL) at 3 time points (pre-intervention, 8 hours after intervention ,and 3-5 weeks post intervention (at the first menstrual cycle after intervention).

Statistical analyses will be conducted by using SPSS 27.0 (IBM Corp.), with a priori power analysis confirming 95% power (α = 0.05; G*Power v3.1.9.7). Data normality will be verified via the Shapiro-Wilk test. Independent Samples t-tests will compare interventional effects between groups, while one-way ANOVA (with LSD post-hoc tests) will analyze multi-point QoL changes. Paired Samples t-tests will evaluate within-group temporal changes (pre vs. post-intervention).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary dysmenorrhea,
* Moderate-to-severe pain during menstrual days 1-3,
* Regular menstrual cycles for past 6 months

Exclusion Criteria:

* Secondary gynaecological conditions,
* Current use of pain medications,
* History of pregnancy

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — As dysmenorrhea is a condition that affects only females so this study will include only females
Enrollment: 46 (Estimated)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) | Before the interventions, after 8 hours from the interventions, & 3-5 weeks post-intervention (first menstrual cycle after interventions)
  It is a pain assessment tool featuring a 10-cm line marked "No pain" (0 cm) and "Worst pain imaginable" (10 cm). Patients indicate their pain level by marking the line, with scores measured in cm (0-10) and categorised as mild (0-3), moderate (4-6), or severe (7-10)

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS-29 Profile v2.0) | Before the interventions, after 8 hours from the interventions, & 3-5 weeks post-intervention (first menstrual cycle after interventions)
  It is a quality of life scale that questions physical function, anxiety, depression, fatigue, sleep disturbance, social roles and activities, pain interference and severity under its subheadings

CONTACTS AND LOCATIONS:
Overall Officials: Gizem Ergezen Şahin, PhD, Study Chair — Medipol University
Locations (1):
- İstanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No